CLINICAL TRIAL: NCT05847829
Title: T-REEX: Phase Locked TRanscranial Electrical EXcitation
Brief Title: Phase Locked TRanscranial Electrical EXcitation
Acronym: T-REEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stichting IMEC-NL (Other)
Collaborators: Stichting Kempenhaeghe (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NL82733.015.22
Record Dates: First submitted 2022-11-25; First posted 2023-05-08 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Novel Method for Transcranial Brain Stimulation
Keywords: Brain stimulation; Closed-loop; Brain activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): The study is open label all participants get the same intervention
  Interventions: Device: T-REEX algorithm

INTERVENTIONS:
Device: T-REEX algorithm — Phase locked transcranial stimulation.

SUMMARY:
Transcranial current stimulation (tCS) has been extensively studied due to its potential of selectively stimulate brain regions in a non-invasive way. However, classic stimulation paradigms are often applied in an open loop configuration, without considering the effects on the underlying brain activity.

Recent studies suggest that when alternating current are used, it would be beneficial to phase lock the stimulation to the target brain wave of interest to achieve selective temporal stimulation, allowing for better control over the stimulation effects.

This study aims at demonstrating a novel setup that allows for precise stimulation targeted in space and time. To achieve that, a combination of tCS and (EEG phased locked) closed-loop modality are used to obtain the required selectivity.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age between 18 and 64

Exclusion Criteria:

* Wounded or particular sensitive skin at areas of investigation. For example, skinrash, discoloration, scars, or open wounds
* Allergies to adhesive or dry electrodes or silver chloride
* Pregnant or lactating
* Any of the following symptoms (fever, tiredness, dry cough, aches and pains, nasal congestion, runny nose, sore throat, diarrhoea)
* Known neurological disorders
* Previous epileptic episodes
* Active implants such as pacemakers or brain stimulators
* Intracranial metal implants

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-10 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
The phase difference (error) between the estimated phase of EEG activity and the phase of the delivered stimulation at the target locationor EEG readout and tCS stimulation | 2 hours

SECONDARY OUTCOMES:
the amount of phase and/or amplitude change in the brain wave of interest (e.g., 10 Hz alpha activity) resulting from different tCS modalities and stimulation parameters used | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Raf van Hoof, PhD, Principal Investigator — Stichting Kempenhaeghe
Locations (1):
- Stichting Kempenhaeghe, Heeze, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No